CLINICAL TRIAL: NCT06222034
Title: An Open-label, Multiple Dose, Multicenter Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Filgotinib in Children and Adolescents From 8 to Less Than 18 Years of Age With Juvenile Idiopathic Arthritis
Brief Title: Study to Measure Filgotinib in the Blood of Children and Teenagers With Arthritis Taking Filgotinib (SCALESIA)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-131; 2023-505844-21-00 (EU CTIS Number)
Record Dates: First submitted 2024-01-04; First posted 2024-01-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Filgotinib Dose A (Experimental): Dose A of filgotinib mini-tablet for participants with bodyweight (BW) 15-<25 kg
  Interventions: Drug: Filgotinib
- Filgotinib Dose B (Experimental): Dose B of filgotinib tablet for participants with BW ≥25-<60 kg
  Interventions: Drug: Filgotinib
- Filgotinib Dose C (Experimental): Dose C of filgotinib tablet for participants with BW ≥60 kg
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Film-coated mini-tablets administered orally once daily
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib Dose A
Drug: Filgotinib — Commercially developed film-coated tablet administered orally once daily
  Other Names: GS-6034; GLPG0634; Jyseleca
  Arms: Filgotinib Dose B; Filgotinib Dose C

SUMMARY:
A Study to evaluate the pharmacokinetics, safety, and tolerability in paediatric population for treating juvenile idiopathic arthritis (JIA).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant with a body mass index (BMI) within the 5th to 95th percentiles for the age and gender (based on World Health Organization BMI charts). Participant must have a minimum weight of 15 kg.
* Participant must meet the International League of Associations for Rheumatology classification for 1 of the following categories and have, according to the investigator's judgment, moderately to severely active disease that is not adequately controlled with his/her current therapy.

  * Rheumatoid factor (RF)-positive polyarthritis
  * RF-negative polyarthritis
  * Oligoarthritis
  * Psoriatic arthritis
  * Enthesis-related arthritis (ERA) Note: Historical Human leukocyte antigen B-27 (HLA-B27) results are considered appropriate for ERA diagnosis during screening.
  * Systemic JIA with active arthritis without active systemic features, or with active systemic features that are stable in the prior 6 months of time of enrollment
* Participant with intolerance or a history of inadequate response to at least one of the following medications for the treatment of JIA, administered for at least 12 weeks, based on current treatment guidelines: conventional synthetic disease-modifying antirheumatic drugs and biological disease-modifying antirheumatic drugs (including methotrexate) and non-steroidal anti-inflammatory drugs for ERA and psoriatic arthritis.
* Female participants of childbearing potential (i.e. who have passed menarche) must have a negative highly sensitive urine pregnancy test.

Key Exclusion Criteria:

* Participant with persistent oligoarthritis.
* Participant with undifferentiated arthritis.
* Participant with any other any other rheumatic, inflammatory, or immunologic disease (e.g. inflammatory bowel disease, hypogammaglobulinemia, systemic lupus erythematosus, or uncontrolled uveitis).
* Active infection that is clinically significant, as per judgment of the investigator.
* Participant with a history of complicated herpes zoster infection (with multi-dermatomal, disseminated, ophthalmic, or central nervous system involvement).
* Currently on any therapy for chronic infection (such as pneumocystis, cytomegalovirus, herpes simplex, or atypical mycobacteria).

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration at steady state of filgotinib (Cmax,ss) | Pre-dose on Day 10, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours post-dose on Day 10
Cmax,ss of GS-829845, major active metabolite | Pre-dose on Day 10, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours post-dose on Day 10
Area under the plasma concentration-time curve over the dosing interval at steady state of filgotinib (AUC0-24,ss) | Pre-dose on Day 10, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours post-dose on Day 10
AUC0-24,ss of GS-829845, major active metabolite | Pre-dose on Day 10, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours post-dose on Day 10
Area under the plasma concentration time curve over the dosing interval at steady state or the effective exposure of filgotinib (AUCeff,ss) | Pre-dose on Day 10, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours post-dose on Day 10
AUCeff,ss of GS-829845, major active metabolite | Pre-dose on Day 10, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 8 hours post-dose on Day 10

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs), TEAEs of interest, serious TEAEs, and TEAEs leading to treatment discontinuation. | Baseline (Day 1) up to week 96
Acceptability of the commercially developed film-coated tablets and of the minitablets as measured by the Pediatric Oral Medicine Acceptability Questionnaire for Patients (POMAQ-P). | Week 4 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Alfasigma Study Director, Study Director — Alfasigma S.p.A.
Locations (10):
- France (2):
  - CHU Amiens - Hopital Nord, Amiens
  - Bicêtre University Hospital, Le Kremlin-Bicêtre
- Germany (3):
  - Children's university hospital Charité, Campus Virchow, SPZ, Berlin
  - Hamburger Zentrum fur Kinder und Jugendrheumatologie, Hamburg
  - Asklepios Klinik Sankt Augustin GmbH, Sankt Augustin
- Malopolskie Badania Kliniczne, Krakow, Poland
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No